CLINICAL TRIAL: NCT06880458
Title: Evaluation of Short-term Changes and Self-reported User Experiences Related to the Know Your OQ™ Initiative
Brief Title: To Validate Changes in Knowledge, Attitudes and Practices (KAPs) Related to the Know Your OQ Initiative and to Understand the Readability, Comprehension and Ease of Use of the Know Your OQ Quiz
Status: Active, not recruiting | Type: Observational
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Other Study IDs: CRO-2024-06 KYOQ-MH
Record Dates: First submitted 2025-01-06; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-01

CONDITIONS: Literacy-language Intervention
Keywords: attitudes; knowledge; oral care
MeSH Terms: conditions — Behavior | interventions — Health Education, Dental

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of Nurses from NAHN: Prospective nurses candidates will be screened to identify those subjects who meet the inclusion/exclusion characteristics. The first 100 subjects who meet the inclusion/exclusion characteristics, sign an Informed Consent Form will be entered into the study.
  Interventions: Other: Oral health education

INTERVENTIONS:
Other: Oral health education — The participants will receive oral health education from multiple different sources, including the Know Your OQ website (https://www.knowyouroq.com/).

SUMMARY:
To validate changes in knowledge, attitudes and practices (KAPs) related to the KnowYour OQ initiative and to understand the readability, comprehension and ease of use of the Know Your OQ quiz

DETAILED DESCRIPTION:
Quantitative analysis will be carried out for changes in knowledge, attitudes and practices(KAPs) after the exposure to the Know Your OQ™ intervention. Qualitative and quantitative analysis will becarried out for readability, comprehension and ease of use of the Know Your OQ™ quiz.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form.
* Male and female subjects aged 18-65+ years old
* Availability for the duration of the study
* English or Spanish fluency
* Access to laptop, tablet or computer with internet/data connection

Exclusion Criteria:

* Not present at NAHn Convention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nurses attending NAHN conference
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-03 (Actual); Primary Completion 2025-07-18 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Knowledge, attitudes and practices towards oral health questionnaire intervention | 1 year
  Once subjects navigate the Know Your OQ webpage, read the provided information on oral health and complete the Know Your OQ survey, they will immediately receive a survey which explores comprehension/readability and general feedback on both the webpage and the Know Your OQ survey. Subjects who indicate negative feedback towards the intervention, including difficulties in understanding the questions of the survey and the material on the webpage, will be invited for a brief follow-up telephone interview and your participation that is optional.

SECONDARY OUTCOMES:
Qualitative Interviews | 1 year
  N=30 nurses who participated in the oral health education intervention and the NAHN community programming will participate in semi-structured qualitative interviews to gain information around oral health practices in their communities, access to oral health care and education, and the community programming.

CONTACTS AND LOCATIONS:
Locations (1):
- National Association of Hispanic Nurses, Lexington, Kentucky, United States